CLINICAL TRIAL: NCT04688268
Title: Find Out the Deciding Factor of Neuromuscular Blocker Dose for Deep Neuromuscular Blockade
Brief Title: Dose for Deep Neuromuscular Blockade Deciding Factor of Neuromuscular Blocker Dose for Deep Neuromuscular Blockade
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, JiWon Han, principal investigator, Seoul National University Bundang Hospital
Other Study IDs: B-2008/633-302
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Laparoscopic Surgery
Keywords: laparoscopic surgery; deep neuromuscular blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- deep neuromuscular blockade: patients who underwent surgery with deep neuromuscular blockade
  Interventions: Drug: deep neuromuscular blockade

INTERVENTIONS:
Drug: deep neuromuscular blockade — Train of Four=0/4, Post tetanic count 1-2

SUMMARY:
Find out the deciding factor(total body weight, corrected body weight, ideal body weight, fat-free mass, body mass index, skeletal muscle mass, body fat) of neuromuscular blocker dose for deep neuromuscular blockade.

DETAILED DESCRIPTION:
Before the surgery, total body weight, corrected body weight, ideal body weight, fat-free mass, body mass index were measured by height and weight and skeletal muscle mass and body fat were measured by Bioelectrical impedance analysis (InbodyH20N). Find the highest correlation between the 8 factors (total body weight, corrected body weight, ideal body weight, fat-free mass, body mass index, skeletal muscle mass, body fat) and the amount of rocuronium administered to deep neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 20-80 and American Society of Anesthesiology Physical Grade (ASA) I-II, who undergo laparoscopic surgery for at least 2 hours under general anesthesia

Exclusion Criteria:

* kidney disease (GFR<60)
* allergy to study drugs
* decline participation
* side effect of propofol and remifentanil
* when anesthesia does not maintain the level of alertness (BIS) below 60 even when the anesthetic dose is increased, or when hemodynamic instability such as bradycardia and hypotension appears

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20-80 and American Society of Anesthesiology Physical Grade (ASA) I-II, who undergo laparoscopic surgery for at least 2 hours under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
the highest correlation coefficient | preoperative 1 days to postoperative 1 days
  the relationship of rocuronium for deep neuromuscular blockade and 8 factors (corrected body weight, ideal body weight, lean body weight, fat-free mass, body mass index, skeletal muscle mass, body fat)

SECONDARY OUTCOMES:
onset time of rocuronium | preoperative 1 days to postoperative 1 days
  time from injection of rocuronium 0.6 mg/kg(TBW) to TOF ratio is less than 0.05
Time to deep neuromuscular blockade | preoperative 1 days to postoperative 1 days
  time from injection of rocuronium 0.6 mg/kg(TBW) to PTC 1
Recovery time | preoperative 1 days to postoperative 1 days
  time from sugammadex injection to TOF ratio > 0.9

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi YJ, Hee Kim Y, Bae GE, Yu JH, Yoon SZ, Kang HW, Lee KS, Kim JH, Lee YS. Relationship between the muscle relaxation effect and body muscle mass measured using bioelectrical impedance analysis: A nonrandomized controlled trial. J Int Med Res. 2019 Apr;47(4):1521-1532. doi: 10.1177/0300060518822197. Epub 2019 Feb 5. PMID 30719949